CLINICAL TRIAL: NCT03701256
Title: Bilateral Transversus Abdominis Plane Block Versus Atracurium During Laparoscopic Gynecology Procedures. Do we Really Still Need the Systemic Neuromuscular Blocking Agents?
Brief Title: Bilateral Transversus Abdominis Plane Block Versus Atracurium During Laparoscopic Gynecology Procedures.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Ben marzouk Sofiene, Professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAP-TRAC
Record Dates: First submitted 2018-10-07; First posted 2018-10-09 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Neuromuscular Blockade; Regional Anesthesia
Keywords: TAP block; curare; laparoscopy; gynecology surgery; abdominal compliance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP Group (Experimental): Bilateral ultrasound TAP bloc performed via 20 ml of 2.5% bupivacaine without neuromuscular blocking agents
  Interventions: Procedure: Bilateral ultrasound guided TAP bloc
- TRAC Group (Active Comparator): Neuromuscular blocking agent: Atracurium 0.1 mg/kg per bolus
  Interventions: Drug: Neuromuscular blockade agent: Atracurium 01mg/kg per bolus

INTERVENTIONS:
Procedure: Bilateral ultrasound guided TAP bloc — In the TAP group: Bilateral ultrasound guided TAP bloc for laparoscopic gynecologic surgery
  Arms: TAP Group
Drug: Neuromuscular blockade agent: Atracurium 01mg/kg per bolus — In the TRAC group: Neuromuscular blockade agent: Atracurium 01mg/kg per bolus for maintaining muscular relaxation and immobilization during laparoscopic gynecologic surgery
  Arms: TRAC Group

SUMMARY:
A monocentric, prospective, randomized controlled trial, including patients proposed for a laparoscopic gynecologic surgery comparing the muscular relaxing effect of a bilateral ultrasound-guided Transversus Abdominis Plane block to usual neuromuscular blockade agent (Atracurium)

DETAILED DESCRIPTION:
We conducted a monocentric randomized single blinded controlled trial for six months starting from February 2015 until July 2015. Patients undergoing laparoscopic gynecologic procedures were included and randomly assigned in two groups receiving either an ultrasound guided TAP block (TAP group) or usual Neuromuscular blockade curare type: Atracurium (TRAC group). Randomization was simple and the allocation sequence was generated by a random number table via computer. The surgeon in charge was blinded about the performance of a TAP block.

Anesthesia protocol was almost the same in the two groups apart from the TAP block performance in the study group and the use of the neuromuscular blockade . No premedication was given to before the procedure. Monitoring was standard with a 5 leads electrocardioscope, non-invasive arterial pressure, pulsed oximetry (SpO2) and pressure of end tidal expired CO2 (PetCO2). Peripheral venous access was obtained and a 0.9 % saline vascular prefilling was done via an 18 or a 16 Gauges (G) percutaneous line in the non-dominant superior member. In the TRAC group, induction was given with 2.5 mg Propofol, 3 γ/kg Fentanyl and 0.6 mg/kg Atracurium. In The TAP group general anesthesia was induced, after a 3 minutes pre-oxygenation, with 3 γ/kg fentanyl, 2.5 mg/kg Propofol and 1mg/kg Suxamethonium. Thereafter the TAP block was performed under ultrasonography guidance with a Samsung (MySonoU6) transportable device and a linear high frequency 5-12 Megahertz transducer. The probe was oriented transversely on the antero-lateral abdominal wall and the image depth was set between 4 and 6 cm. Once anatomic structures were visualized and well distinct, the probe was moved posteriorly until the mid-axillary line between the 12th rib and the iliac crest. Operator should be able to identify from top to bottom: the subcutaneous fat tissue (hypo-echogenic), External Oblic Abdominal Muscle (EOAM), Internal Oblic Abdominal Muscle (IOAM), Transverse Abdominis Muscle (TAM) (heterogeneous), peritoneum (hyper-echogenic) and underneath intraabdominal organs both moving with respiration. The junction between the posterior fascia of the IOAM and the anterior fascia of the TAM is also hyper-echogenic and represent the region of interest as it is the local anesthetic injection site. The puncture was proceeded with 100 mm lenght needle 21 G (Vygon, France) needle witch progressed obliquely through the abdominal wall. Operator realized an in plane ultrasound guided approach. As soon as the tip of the needle was placed in the junction between the IOAM and TAM and the aspiration test negative, a priming of 3 ml local anesthetic injection was used in order to unsure a correct position of the needle. In this case the injectate would appear as a hypo-echogenic oval well-shaped volume spreading between the two muscle layers. An inaccurate injection was suspected by the absence of the described image. Intramuscular injection could appear as a poorly defined hyper-echogenic image within the muscle. Once the correct position verified, the rest of the 20 ml of the 2.5% bupivacaine is injected. The contralateral block was performed equally. Anesthesia was maintained by a total intravenous anesthesia in both groups. Fentanyl was systematically reinjected every 30 minutes and Propofol was infused at 8-10 mg/kg/h. In the TRAC group, Atracurium reinjections were guided by the monitoring of the NMB every 20 minute at a dose equal to 0.1mg/kg to be reevaluated after 5 minutes. In the TAP group, a rescue injection of NMB agent was indicated in case of diaphragmatic contractions, surgeons' complaint or patients' movement after optimization of narcosis by increasing propofol infusing speed to a maximum of 5 mg/kg/h beyond the baseline speed and checking analgesia. In both groups patients were ventilated on a volume assisted mode with 50 % of inspired fraction of Oxygen and 4-6 cmH2O of positive end expiratory pressure (PEEP) aiming to get an SpO2>95%. Tidal volume and respiratory rate were set as to maintain a PetCO2 between 30 and 45 mmHg. A nasogastric tube was inserted before trocars introduction (T0). Patients from the two study groups had a postoperative analgesia prescription including acetaminophen (1g/6h), Ketoprofen (100 mg/12h) and Nefopam (20mg/4h). A 5 mg subcutaneous morphine injection was considered as rescue analgesia.

ELIGIBILITY:
Inclusion Criteria:

* American Association of anesthesiologists' class I to III (ASA I to ASA III)
* undergoing laparoscopic gynecologic procedures

Non inclusion Criteria:

* patients' refusal to be part of the study
* ASA IV and higher
* known allergic history to Propofol or any of its components (eggs, soya and beans, etc.), suxamethonium, Fentanyl or Atracurium.
* Patients who presents any regional anesthesia contraindication as clotting disorders, injection site infection and allergy to local anesthetics
* Psychiatric and neurologic disorders and the inability to understand pain scores and the study protocol

Exclusion Criteria:

* unsuccessful TAP block
* Observed anesthesia or surgical incident which requires the end of the ongoing procedure or the conversion to laparotomy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2015-10-31 (Actual)

PRIMARY OUTCOMES:
Abdominal compliance (Ca) | peroperatively every 10 minute from the introduction of the laparoscopy trocars until their removal
  Ca calculation was based on the formula: Ca= ΔV/ΔP with ΔV and ΔP referring to the volume variation of CO2 insufflated and ΔP to the variation of intraabdominal pressure during the procedure
surgeon satisfaction | peroperatively
  Surgeons were asked at the end of the procedure about their satisfaction. Their answers were put on a scale between 1 and 4 (1: poor, 2: average, 3: good, 4: excellent)

SECONDARY OUTCOMES:
Heart Rate (HR) (bpm) | peropertively from the laparoscopy trocars introduction until skin closure
  Heart rate
Mean arterial pressure (MAP) (mmHg) | peropertively from the laparoscopy trocars introduction until skin closure
  Mean arterial pressure
SpO2 (%) | peropertively from the laparoscopy trocars introduction until skin closure
  pulsed oxygen saturation
PetCO2 (mmHg) | peropertively from the laparoscopy trocars introduction until skin closure
  End Tidal CO2 pressure
Pp (cmH2O) | peopertively from the laparoscopy trocars introduction until skin closure
  Plateau pressure
awakening time after disruption/discontinuing analgesia | peropertaively
  time needed for extubation after discontinuing anesthesia maintenance
diaphgram mouvement | peropertively
  diphgram mouvement assessed on the ventilator or in the laparoscopy monitor
surgeons complaint | peropertaively
  surgeons complaints about operation conditions

CONTACTS AND LOCATIONS:
Overall Officials: Hayen Maghrebi, Professor, Study Chair — Tunis Maternity Center
Locations (1):
- Tunis maternity and neonatology center,, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided